CLINICAL TRIAL: NCT00286052
Title: The Impact of Concomitant Ultra Low Dose Infusion Naloxone and Therapeutic Infusion Opioid on Opioid Requirements in Pediatric ICU Patients
Brief Title: Impact of Low Dose Naloxone on Fentanyl Requirements in Pediatric ICU Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB File: 1002-605
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2005-09

CONDITIONS: Opioid Tolerance
MeSH Terms: interventions — Naloxone

INTERVENTIONS:
Drug: Low Dose Naloxone

SUMMARY:
Recently there has been an increased awareness in the need for adequate sedation and pain control for Pediatric Intensive Care Unit (ICU) patients. Fentanyl is an opioid commonly used in Pediatric ICU patients to decrease pain and increase sedation. Although opioids (e.g. morphine and fentanyl) provide excellent pain relief, they have many side effects including dependence, tolerance and withdrawal. These side effects lead to increased doses in order to maintain pain control and/or sedation. There have been a few adult studies pointing to some possible treatments. For example, giving low dose naloxone along with opioids. Adult studies show that this combination not only decreases the frequency of opioid side effects, but also improves pain control and prevents the development of tolerance. We propose that children who receive low dose naloxone infusions along with fentanyl infusions will demonstrate: 1) decreased total daily doses of Fentanyl, 2) decreased frequency of withdrawal and 3) increased pain and sedation control. In this randomized, blinded prospective trial we will enroll 168 Pediatric ICU patients. Patients will receive either low dose naloxone or placebo simultaneously with their fentanyl infusion. Pain and sedation will be assessed using the Modified Motor Activity Assessment Scale (MMAAS). The fentanyl infusion will be increased to provide adequate pain control and/or sedation. Naloxone infusion will not be adjusted. Approximately 48 hours prior to removal from the ventilator, patients will have their fentanyl infusions decreased while being monitored for withdrawal. Patients showing signs of withdrawal will receive methadone, an opioid taken by mouth. Once off fentanyl, naloxone will be stopped. Patients will continue to be monitored for withdrawal for 4 days or until ICU discharge. If this study works, patients who receive low dose naloxone along with opioid infusions will have less tolerance and dependence and demonstrate less withdrawal. This may cause shorter Intensive Care Unit stays.

DETAILED DESCRIPTION:
Objective:

To determine if Naloxone administration to pediatric ICU patients on Fentanyl infusions require less Fentanyl compared to control patients.

Background:

During recent years there has been an increased awareness of the need for adequate sedation and analgesia of critically ill pediatric patients. The choices of the treatment of pain are numerous, but in the Pediatric ICU parenteral opioids are most commonly used. At equipotent doses, all mu agonist opioids (Morphine, Fentanyl, Meperidine and Codeine) produce similar physiologic effects and side effects. Opioids can cause hypoventilation, hypotension, constipation and cause urinary retention. Patients receiving continuous opioid infusions experience not only these physiologic side effects, but also the side effects of dependence, tolerance and withdrawal. These last side effects complicate medical issues and contribute to longer ICU admissions.

Anand wrote a review article addressing the problems of drug dependence and withdrawal in the PICU. In his article he discussed the mechanisms, pharmacology and presentation of opioid withdrawal. He also discussed prevention of opioid withdrawal including such therapies as the concomitant infusion of opioid agonists and low dose Naloxone. Tobias also wrote a review article describing the consequences of the prolonged use of sedative and analgesic agents in the Pediatric ICU. Among the problems of note are tolerance, dependence and withdrawal in the Pediatric ICU. He discussed several possible therapies for the treatment and prevention of opioid withdrawal. Among these was the concomitant infusion of opioid agonist and low dose Naloxone, an opioid agonist. Naloxone selectively blocks those opioid receptors that are coupled with stimulatory G proteins, thus blocking mechanisms for super-activation of the cAMP pathway. This improves the efficacy of analgesia and prevents the development of acute tolerance.

Recent preclinical and clinical studies (Crain, Gan, Levine, Joshi) have shown that co-treatments with extremely low doses of opioid receptor antagonists can markedly enhance the efficacy specific to Morphine and related analgesics. Crain did studies using Naloxone, in-vitro and in-vivo, that show direct competitive antagonism of Gs coupled excitatory opioid receptor functions. This markedly enhances Morphine's antinociceptive potency and simultaneously attenuates opioid tolerance and dependence.

Studies by Gan and Levine with adult post-op hysterectomy patients in one study and adult patients following tooth extraction in a separate study show that low dose Naloxone could enhance the analgesic potency of opioid agonists. The striking consistency of these studies provides evidence that clinical treatment of pain can be improved by administering opioid analgesics together with low doses of excitatory opioid receptor antagonists. The possibility of these same effects occurring in Pediatric ICU patients has not been explored.

Hypothesis:

Children admitted to the Pediatric ICU requiring continuous infusions of opioids who receive low dose Naloxone infusions will have a 30% decrease in the maximum total daily dose of Fentanyl and a decreased need for escalating doses of continuous infusions during ICU admission.

Study Design:

This will be a prospective double-blinded randomized placebo-controlled study. Patients admitted to the ICU and consented for the study will be started on either Naloxone continuous infusion of 0.25micrograms/kilogram/hour (mcg/kg/hr) or normal saline continuous infusion at equal rate and volume to be determined by the pharmacy. The dose or rate of Naloxone infusion will not be manipulated throughout the study.

During the first four hours of ICU admission the patients will be assessed hourly via the Modified Motor Activity Assessment Scale (MMAAS, see appendix 1). Adjustments will be made to Fentanyl and Midazolam infusions according to protocol for patients not achieving a sedation score of -1 to +1 (see figure 1). Patients with score of greater than +1 and associated tachycardia/hypertension will receive a bolus of Fentanyl and repeat MMAAS in 30 minutes. The Fentanyl bolus will be equal to one hour total dose of Fentanyl infusion with considerations for weight. Dosage will be adjusted for weight accordingly: 1mcg/kg for children less than 50kg and 0.5mcg/kg for children greater than 50kg. If repeat MMAAS score is again greater than +1 with hypertension/tachycardia the patient will receive another bolus of Fentanyl (dose as denoted above) and will have increase of Fentanyl infusion by 1mcg/kg/hr. The patient will have repeat MMAAS 30 minutes after change. If repeat MMAAS score still greater than +1 a physician will be called for assessment and intervention. If the first repeat MMAAS score is greater than +1 with no hypertension/tachycardia the patient will receive a bolus of Midazolam. The Midazolam bolus will be either equal to one hour total dose of Midazolam infusion or 0.1mg/kg with considerations for weight. Dosage will be adjusted according for weight: 0.1mg/kg for children less than 20kg or 0.05mg/kg for children greater than 20kg. The patient will have repeat MMAAS in 30 minutes. If second MMAAS score still greater than +1 a physician will be called for assessment and intervention. If MMAAS score at any time between +1 and -1 then repeat MMAAS will be repeated at next scheduled time per protocol (see figure 2).

If patients require an increase of more than 2 mcg/kg/hr within 3 hours, then the patient will have Midazolam either started or increased. Dosage will be 0.1 mg/kg/hr for children less than 20kg and 0.05 mg/kg/hr for children over 20kg for starting Midazolam. Dosage for increase in current infusion will be 0.1mg/kg/hr for children less than 20kg and 0.05mg/kg/hr for children over 20kg.

Patients will be assessed hourly, using the MMAAS, for the first four hours of admission to the study and then every 2 hours for the subsequent 8 hours. After this initial time period patients will be assessed every 4 hours until completion of the study. Each assessment will consist of recording the sedation score, temperature, heart rate, respiratory rate, ventilator set rate, blood pressure, oxygen saturation, infusion rate of Fentanyl and/or Midazolam and the need for any intervention and what that intervention included. Patients with signs of increased pain/discomfort will be assessed using the sedation scale as needed between scheduled assessments. Interventions will be made per protocol as needed between scheduled assessments. Once pt MMAAS score between +1 and -1 the patient will resume scheduled MMAAS evaluations according to protocol.

If the patient has a sedation score of <-1 on MMAAS, among any of the scheduled or intermittent assessments, the Midazolam infusion will be decreased by 0.05 mg/kg/hr and the patient will be reassessed in two hours. If there is no Midazolam infusion then, the Fentanyl infusion will be decreased by 0.5mcg/kg/hr and the patient will be reassessed in two hours. If the patient continues to have pain score of <-1 on repeat MMAAS then the Fentanyl or Midazolam continuous infusion will again be decreased as denoted above. The patient will again be reassessed in two hours. If the patient continues to have MMAAS score of <-1 a physician will be notified for assessment and intervention. If repeat MMAAS score >+1 then Fentanyl infusion will be increased and noted above and the patient will be reassessed in 30 min. If second repeat MMAAS not between +1 and -1 then a physician will be notified for assessment and intervention. If at any time MMAAS score between +1 and -1 then MMAAS will be repeated per protocol. If following first decrease in infusion and repeat MMAAS score >+1 then infusion previous adjusted will be increased to prior dose. The patient will be reassessed in 30 minutes. If repeat MMAAS score >+1 with hypertension/tachycardia then Fentanyl infusion will be increased as noted above. If MMAAS score >+1 and not hypertension/tachycardia then Midazolam infusion will be increases as noted above. After intervention MMAAS will be repeated in 30 minutes. If repeat MMAAS score remains >+1 then a physician will be notified for assessment and intervention (see figure 3).

As the patients approach 48-72 hours near the end of the need for continuous infusion or opioid, per decision by the medical staff, they will be weaned from infusions. The Naloxone infusion will remain unchanged. The Naloxone infusion or normal saline infusion will be discontinued when the Fentanyl infusion is discontinued. The Fentanyl infusions will be decreased by 25% of original dose every 12 hours until off. Once patients start the Fentanyl wean they will have withdrawal assessed every six hours and as needed using the Modified Narcotic Withdrawal Scale (MNAS, see appendix 2). Patients receiving two successive scores of 8 or above will be determined to have withdrawal. These patients will be started on Methadone as directed by the primary team and Fentanyl infusion will continue to be decreased by 25% every 12 hours until off. As patients are weaned from continuous infusions they will continue to have assessments every 6 hours using MNAS until infusions are discontinued. Once the continuous infusion of Fentanyl is discontinued the patient information will continue to be monitored using MNAS and vital signs stated earlier for 4 days or until ICU discharge.

Any need for reinstitution of continuous infusion of Fentanyl and the medical reason for such action will be noted. Increases in oral agents after receiving the first four doses will be noted. The need for intermittent boluses of IV analgesia or sedation during the weaning and associated medical reasons will be noted. These things will be monitored for the duration of the study.

Patients may receive bolus of any medication as ordered by physicians for procedures without interfering with the study. Notation of such action will be made with next assessment. If at any time a physician deems it necessary to begin a medication not classified as an opioid or benzodiazepine the patient will be removed from the study. If at any time a physician begins a scheduled dose of an additional opioid or benzodiazepine to total more than one of each class the patient will be removed from the study.

Adverse events (nausea, vomiting, sweating, tachycardia, increased blood pressure, tremulousness, seizures and cardiac arrest) will be noted in the medical record. If medical reasons for such events are ruled out then the patient will be unblinded from the study.

Statistical Analysis An SPSS software random number generator was used to create a permuted block randomization schedule. Patient assignment was unknown to all investigators and medical team members, with the exception of the PICU pharmacist.

Power analysis was based upon an assumed power of 80%, an effect size of 30% reduction in maximum cumulative daily dose of fentanyl, and historical data for maximum daily fentanyl dosing in the PICU at Children's Medical Center Dallas (Between January and August 2002, the cumulative maximum daily fentanyl dose of 428 PICU patients was 79 mcg/kg with a standard deviation of ± 47 mcg/kg). Thus, the sample size was determined to be 62 per group (total N=124). The alpha criterion for significance was considered 0.05.

All parametric and nonparametric data were analyzed using SPSS for Windows and Microsoft Excel software packages. Interim monitoring at the midpoint of the study was performed by an independent Data and Safety Monitoring Board (DSMB), which consisted of both internal and external reviewers. O'Brien-Fleming stopping boundaries and Lan-DeMets spending functions were employed in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children age one (1) day to eighteen (18) years, requiring admission to the Pediatric ICU, requiring continuous infusion of Fentanyl analgesic anticipated to last greater than 4 days will be eligible for enrollment. Patients from both genders, all races and ethnic backgrounds will be eligible. Patients meeting the above criteria will be eligible regardless of nutritional status, performance status or recovery from prior medical treatment. They will not be excluded if they require simultaneous infusions of sedation with Midazolam. Enrollment will require parental consent.

Exclusion Criteria:

* Patients will not be eligible if they meet any of the following criteria:
* Patients who are currently on oral analgesia or sedation
* Patients who have a prior history of drug or alcohol dependence/abuse.
* History of significant or preexisting cardiovascular disease, they are receiving pro-arrhythmia medications, such as class I, II, III or IV antiarrhythmic agents.
* Patients who are allergic to opioids or opioid antagonists.
* Patients with documented chromosomal abnormality impairing perception of pain/discomfort.
* Unable to obtain parental or legal guardian's informed consent
* Concurrent admission to another study.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 128
Dates: Start 2002-12; Study Completion 2004-08

PRIMARY OUTCOMES:
Maximum Cummulative Daily Fentanyl Dose

SECONDARY OUTCOMES:
Number of Rescue Fentanyl Boluses
Number of Rescue Midazolam Boluses
Total Midazolam Dose
Narcotic Withdrawal Scale Score
Modified Motor Activity Assessment Score

CONTACTS AND LOCATIONS:
Overall Officials: Cindy M Darnell, Principal Investigator — University of Texas
Locations (1):
- Unversity of Texas Southwestern, Children's Medical Center, Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Darnell CM, Thompson J, Stromberg D, Roy L, Sheeran P. Effect of low-dose naloxone infusion on fentanyl requirements in critically ill children. Pediatrics. 2008 May;121(5):e1363-71. doi: 10.1542/peds.2007-1468. Epub 2008 Apr 14. PMID 18411237